CLINICAL TRIAL: NCT04983849
Title: Evaluation of Effects of Subgingival Administration of Metronidazole Hydrogel 25% in Stage II and III Periodontitis: Randomized, Split Mouth, Single-blind Trial.
Brief Title: Evaluation of Metronidazole Hydrogel 25% in Stage II and III Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of L'Aquila (Other)
Responsible Party: Principal Investigator, Enrico Marchetti, Prof. Enrico Marchetti, University of L'Aquila
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Prot. RCT 001/2021
Record Dates: First submitted 2021-07-20; First posted 2021-07-30 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Periodontitis
Keywords: Periodontitis; Periodontal disease
MeSH Terms: conditions — Periodontitis; Periodontal Diseases | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hydrogel metronidazole 25% (Active Comparator): metronidazole hydrogel in adjunct to non surgical periodontal therapy
  Interventions: Drug: metronidazole hydrogel
- scaling and root planing (Active Comparator): the only use of scaling and root planing
  Interventions: Procedure: scaling and root planning

INTERVENTIONS:
Drug: metronidazole hydrogel — scaling and root planning in adjunct to the use of metronidazole in the periodontal pocket
  Other Names: Non Surgical Periodontal Therapy
  Arms: hydrogel metronidazole 25%
Procedure: scaling and root planning — scaling and root planning
  Arms: scaling and root planing

SUMMARY:
A randomized clinical trial will be performed single-blind to evaluate the effectiveness of sublingual metronidazole hydrogel 25 % in periodontitis.

DETAILED DESCRIPTION:
A randomized clinical trial will be performed single-blind to evaluate the effectiveness of sublingual metronidazole hydrogel 25 % in periodontitis in stage II and III.

At least 40 volunteers between the age of 18 and 80, will be enlisted, with the need to perform the SRP. In half of the mouth will be used the metronidazole hydrogel 25%, while in the other half no drugs will be used of delivered.

The study will be carried out in accordance with the Helsinki Declaration and the Protocol will be submitted to the Internal Review Board of the University to obtain authorization. Afterwards, the protocol will be recorded on the databa-se clinicaltrials.gov for clinical trials.

The protocol respects the SPIRIT parameters for the compilation of protocols on clinical trials and the study will respect the parameters of CONSORT sta-tement on randomized clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* 10% of sites with survey depth 5 mm
* Comparable pockets in 4 mouth quadrants
* Health at systemic level

Exclusion Criteria:

* Changes in oral mucosa
* Depth at the poll 5 mm
* Presence of removable prostheses or orthodontic equipment
* Allergies to even a single component of a product in testing• Antibiotic-based treatments during the 6 months preceding the start of testing
* History of previous periodontal treatments in the 12 months preceding the start of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Concentration of MMP8 | baseline - 1 week
  matrix metalloproteinases (ng/ml)
Concentration of MMP9 | baseline - 1 week
  matrix metalloproteinases (ng/ml)
Concentration of IL1 | baseline - 1 week
  interleukin (pg/ml)
Concentration of IL6 | baseline - 1 week
  interleukin (pg/ml)
Concentration of IL8 | baseline - 1 week
  interleukin (pg/ml)
Concentration of IL17 | baseline - 1 week
  interleukin (pg/ml)
Concentration of TNF alfa | baseline - 1 week
  tumor necrosis factor alfa (pg/ml)
Concentration of RANK-L | baseline - 1 week
  Receptor activator of nuclear factor kappa-Β ligand (pg/ml)
Concentration of OPG | baseline - 1 week
  osteoprotegerin (pg/ml)

SECONDARY OUTCOMES:
CAL | baseline - 1 week
  clinical attack level (mm)
PPD | baseline - 1 week
  Probing Pocket Depth (mm)
GI | baseline - 1 week
  gingival index (0-3)
FMPS | baseline - 1 week
  full mouth plaque score (0-100%)
FMBS | baseline - 1 week
  full mouth bleeding score (0-100%)

CONTACTS AND LOCATIONS:
Locations (1):
- University of L'Aquila, division of periodontology, L’Aquila, Italy

IPD SHARING:
Plan to Share IPD: Undecided